CLINICAL TRIAL: NCT03738488
Title: 3D-biomodels for Surgical Planning in Patients With Renal Cancer and Vascular Involvement
Acronym: 3DUrologia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundación Pública Andaluza para la gestión de la Investigación en Sevilla (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: Trials 3D Urologia
Record Dates: First submitted 2018-10-18; First posted 2018-11-13 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: Renal Cell Carcinoma; Three-Dimensional; Venous Thromboses
MeSH Terms: conditions — Carcinoma, Renal Cell; Venous Thrombosis | interventions — Imaging, Three-Dimensional

STUDY DESIGN:
Intervention Model Description: Study model: Longitudinal, prospective, experimental, multi centric on a cohort of patients diagnosed of Renal Cell Carcinoma with Vascular Involvement from 2018 in either the HUVR or the HURC
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D printing + images (Experimental): Surgery planification with the combination of all the images available and a 3D biomodel printed from that images.
  Interventions: Device: 3D printing + images
- Images (Active Comparator): Surgery planification with all the images available
  Interventions: Other: Images

INTERVENTIONS:
Device: 3D printing + images — To perform a surgery planification with the combination of the images available and the 3D biomodel in terms of: anticipation of potential complications and the human resources and necessary materials
  Arms: 3D printing + images
Other: Images — To perform a surgery planification with the images available in terms of: anticipation of potential complications and the human resources and necessary materials
  Arms: Images

SUMMARY:
Objectives:

Apply 3D- printed biomodels in patients with renal cancer (RCa) and vascular involvement (VTT) to: (1) improve surgical planning, (2) upgrade surgical results, (3) facilitate communication with patients, (4) serve as a model for teaching residents and (5) shortening the learning curve in experienced urologists.

Methodology:

The design of the study is a randomized clinical trial, to determine the safety, precision, feasibility, predictability, efficacy and efficiency of a surgical strategy based on imaging tests and 3D models regarding the surgical planning in patients with RCa and VTT. This is a longitudinal, prospective, experimental and multicenter study on a cohort diagnosed of RCa and VTT from 2018 in the Virgen del Rocío University Hospital (HUVR) or in the Ramón y Cajal University Hospital (HURC). The study will last for 3 years and will be carried out jointly by the HUVR, the HURC and the IBIS, in a multidisciplinary team made up of urologists, radiologists and engineers.

DETAILED DESCRIPTION:
Phase 1, obtaining the 3D printed biomodel and study of feasibility.

Distribution of tasks: Conducted jointly by:

* Radiology team of the HUVR: Segmentation and 3D virtual reconstruction of the image tests. Compare measurements with image tests.
* IBIS / HUVR engineering team. Design and development of specific segmentation algorithm for the tissue selection of interest. Modeling of image and printing of the 3D model.
* Urology team of the HUVR. Identification of anatomical structures and taking measurements in the 3D model. Simulation of surgery following the surgical guide.
* Production center: It will be carried out entirely in the HUVR.
* Process: custom and manufacture 3D models to perform a surgical simulation using imaging tests of operated patients, with different characteristics until achieving an optimum prototype. Different anatomical structures will be measured and compared in the model and in the image (Collection sheet of data). Later, we will check if it is possible to perform a surgical simulation on the model reproducing in it each of the steps necessary to perform the surgery (surgical guide, annex 3).

Phase 2, precision and predictability study:

Distribution of tasks: Conducted jointly by:

* HUVR radiology team and HURC radiology team. Segmentation and 3D virtual reconstruction of the image tests. Taking measurements in image tests.
* IBIS / HUVR engineering team. 3D model printing.
* HUVR urology team and urology team HURC. Taking measurements in the 3D model. Surgical planning with imaging tests or with imaging tests and 3D model (simulation following the surgical guide).

Real surgery and taking measurements in real surgery.

* Production center: 3D printing in the HUVR, precision and predictability study, HUVR and HURC.
* Process: all patients diagnosed with CaR and TTV in the HUVR and HURC will be recruited between the years 2018 and 2021 and will be randomized into two groups. In the control group the surgical planning will be based exclusively on image tests. In the intervention group we will carry out a surgical planning based on imaging tests and the 3D model (on which we will perform a surgical simulation following the guide surgical). Subsequently, the surgery will be carried out, and in each of the groups it will be compared (Gold Standard) with the pre-surgical planning performed.
* precision study Anatomical measurements will be taken before the surgical intervention in the image models, in the 3D model and subsequently in vivo during surgery
* predictability study A prediction will be made of the type of surgery to be performed, the complications, and the necessary human and material resources.

Phase 3, efficacy and efficiency study:

* HUVR urology team and urology team HURC. Data Collect.
* Process: We will check if a surgical planning with image tests and 3D model makes the surgery more effective and efficient than the one based exclusively on imaging tests. Efficacy, will be defined as the ability to achieve a good surgical result. Efficiency will be defined as the ability to obtain good results with the minimum possible costs and in the minimum possible time.

Phase 4, study of satisfaction level with surgical planning based on 3D model and learning curve of urologists:

* HUVR Urology team and HURC urology team: Delivery of satisfaction surveys and data collection.
* HUVR urology team: Comparison of learning curves.

Final phase, analysis of the results and dissemination plan.

- All researchers: the results of the different tasks carried out in the project will be evaluated and scientific publications and communications in national and international congresses will be made.

ELIGIBILITY:
Inclusion Criteria:

* Signature of informed consent.
* Age over 18 years or between 14 and 18 with the authorization from mother / father / guardian.
* Diagnosed of renal cancer with vascular involvement in the HUVR or HURC between 2018 and 2021

Exclusion Criteria:

* Pregnant.
* Immunosuppression.
* No signature of informed consent.
* Impossibility of monitoring or follow up.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2019-12-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-05-30 (Estimated)

PRIMARY OUTCOMES:
Grade of Concordance between the CT and the 3D model evaluated with the kappa and the intraclass correlation coefficient. | 12 weeks, from the beginning of the study and before recruitment starts
  The grade of concordance between the CT and 3D model will be assessed firstly identifying all the anatomical structures in the 3D model: Kidneys, tumor, arteries and veins.Then some measures will be taken both in the CT and the model to compare them. That will be repeated in 20 cases and the grade of concordance will be assessed by using the Kappa and the intraclass correlation coefficient.

SECONDARY OUTCOMES:
Grade of concordance between the CT and/or 3D model and the vivo model evaluated with the kappa and the intraclass correlation coefficient. | 1 year, since the recruitment begins until we have the first 10 cases of renal cell carcinoma with thrombus venous extension operated
  The grade of concordance between the CT and/or 3D model and the "vivo" will be assessed firstly identifying all the anatomical structures in the CT or 3D and the vivo when the surgery is performed: Kidneys, tumor, arteries and veins.Then some measures will be taken both in the CT and or 3D and the vivo during the surgery to compare them. The grade of concordance will be assessed by using the Kappa and the intraclass correlation coefficient.
Grade of predictability of the surgery planning with 3D and images compared with the surgery planning made only with images. It will be assessed by using the Kappa and the intraclass correlation coefficient. | 3 years, since the recruitment begins until the end of the recruitment.
  A pre-surgery planning will be made to predict the kind of surgery, the potential complications and the human and material necessary resources for the surgery. Both predictions (the one made only with images, and the one made with images and 3D) will be compared with the reality (the surgery). The grade of concordance between the prediction and the reality will be assessed using the Kappa and the intraclass correlation coefficient.
Surgery outcome in terms of blood transfusion (number of blood transfusions needed) | 3 years, since the recruitment begins until the end of the recruitment.
  We will compare the surgery outcomes between the surgery pre-planned with images and the one pre-planned with 3D and images. That will be assessed in terms of blood transfusion (number of blood transfusiones needed)
Surgery outcome in terms of number and grade of complications according to Clavien's scale | 3 years, since the recruitment begins until the end of the recruitment.
  We will compare the surgery outcomes between the surgery pre-planned with images and the one pre-planned with 3D and images. That will be assessed in terms of number and grade of complications following the Clavien's scale.
Surgery outcome in terms of free surgery margins according to the histopathology analysis of the specimen. | 3 years, since the recruitment begins until the end of the recruitment.
  We will compare the surgery outcomes between the surgery pre-planned with images and the one pre-planned with 3D and images. That will be assessed in terms of free surgery margins according to the histopathology analysis of the specimen (yes/no)
Surgery outcome in terms of number of hospitalisation days | 3 years, since the recruitment begins until the end of the recruitment.
  We will compare the surgery outcomes between the surgery pre-planned with images and the one pre-planned with 3D and images. That will be assessed in terms of number of hospitalisation days
Surgery outcome in terms of necessity of stay in the Intensive Care Unit | 3 years, since the recruitment begins until the end of the recruitment.
  We will compare the surgery outcomes between the surgery pre-planned with images and the one pre-planned with 3D and images. That will be assessed in terms of necessity of stay in the Intensive Care Unit (yes/no)
Cost-effectiveness analysis, comparing the cost of the surgery with the 3D planning and the image planning. | 3 years, after the recruitment is ended
  Cost-effectiveness analysis, comparing the cost of the surgery with the 3D planning (sum of the impression, the surgery and the postoperative time) and the surgery performed with an image planning.
Comparison of learning curves using the CUSUM method. | 3 years, after the recruitment is ended and all the surgeries performed
  We will compare the learning curve of the surgeon that starts its training practicing in a 3D model and the one of a surgeon that did the learning curve without training in the 3D model
Satisfaction level, assessed by a specifically designed questionnaire to evaluate the satisfaction with the 3D model of both urologists and patients (questionnaire published in DOI 10.1007/s00345-015-1632-2 and https://doi.org/10.1007/s00345-017-2126-1) | 3 years. The satisfaction questionnaire to the patient will be given in the consult that the surgery is explained with the 3D model. At the end of the study, after the third year the satisfaction questionnaire will be given to all the urologists.
  A questionnaire will be given to each patient in the consult after the explanation of the surgery with the 3D model (2 questionnaire published in DOI 10.1007/s00345-015-1632-2) In addition, at the end of the study, another satisfaction questionnaire will be given to all the urologists that participated in the study using a questionnaire already used (https://doi.org/10.1007/s00345-017-2126-1)

CONTACTS AND LOCATIONS:
Overall Officials: Carmen Belén Congregado Ruíz, FEA, Principal Investigator — Virgen del Rocío University Hospital
Locations (2):
- Spain (2):
  - Ramón y Cajal University Hospital, Madrid
  - Virgen del Rocio University Hospital, Seville

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication will be shared, as well as the study protocol, the Statistical Analysis Plan, the Informed Consent Form and the Clinical Study Report
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Starting on november 2018 until may 2022
Access Criteria: IPD and any additional supporting information will be shared, with any physician interested in the protocol, the biomodel the Statistical Analysis or the clinical study report. This information will be given always without revealing the identity of the participants of the study

REFERENCES:
- [Background] Gupta K, Miller JD, Li JZ, Russell MW, Charbonneau C. Epidemiologic and socioeconomic burden of metastatic renal cell carcinoma (mRCC): a literature review. Cancer Treat Rev. 2008 May;34(3):193-205. doi: 10.1016/j.ctrv.2007.12.001. Epub 2008 Mar 4. PMID 18313224
- [Background] Knoedler M, Feibus AH, Lange A, Maddox MM, Ledet E, Thomas R, Silberstein JL. Individualized Physical 3-dimensional Kidney Tumor Models Constructed From 3-dimensional Printers Result in Improved Trainee Anatomic Understanding. Urology. 2015 Jun;85(6):1257-61. doi: 10.1016/j.urology.2015.02.053. PMID 26099870
- [Background] Hatakeyama S, Yoneyama T, Hamano I, Murasawa H, Narita T, Oikawa M, Hagiwara K, Noro D, Tanaka T, Tanaka Y, Hashimoto Y, Koie T, Ohyama C. Prognostic benefit of surgical management in renal cell carcinoma patients with thrombus extending to the renal vein and inferior vena cava: 17-year experience at a single center. BMC Urol. 2013 Oct 14;13:47. doi: 10.1186/1471-2490-13-47. PMID 24125174
- [Background] Bissada NK, Yakout HH, Babanouri A, Elsalamony T, Fahmy W, Gunham M, Hull GW, Chaudhary UB. Long-term experience with management of renal cell carcinoma involving the inferior vena cava. Urology. 2003 Jan;61(1):89-92. doi: 10.1016/s0090-4295(02)02119-2. PMID 12559273
- [Background] Blute ML, Boorjian SA, Leibovich BC, Lohse CM, Frank I, Karnes RJ. Results of inferior vena caval interruption by greenfield filter, ligation or resection during radical nephrectomy and tumor thrombectomy. J Urol. 2007 Aug;178(2):440-5; discussion 444. doi: 10.1016/j.juro.2007.03.121. Epub 2007 Jun 11. PMID 17561151
- [Background] Craven WM, Redmond PL, Kumpe DA, Durham JD, Wettlaufer JN. Planned delayed nephrectomy after ethanol embolization of renal carcinoma. J Urol. 1991 Sep;146(3):704-8. doi: 10.1016/s0022-5347(17)37899-0. PMID 1875477
- [Background] Psutka SP, Boorjian SA, Thompson RH, Schmit GD, Schmitz JJ, Bower TC, Stewart SB, Lohse CM, Cheville JC, Leibovich BC. Clinical and radiographic predictors of the need for inferior vena cava resection during nephrectomy for patients with renal cell carcinoma and caval tumour thrombus. BJU Int. 2015 Sep;116(3):388-96. doi: 10.1111/bju.13005. Epub 2015 Mar 23. PMID 25430786
- [Background] D'Urso PS, Barker TM, Earwaker WJ, Bruce LJ, Atkinson RL, Lanigan MW, Arvier JF, Effeney DJ. Stereolithographic biomodelling in cranio-maxillofacial surgery: a prospective trial. J Craniomaxillofac Surg. 1999 Feb;27(1):30-7. doi: 10.1016/s1010-5182(99)80007-9. PMID 10188125
- [Background] Levine JP, Patel A, Saadeh PB, Hirsch DL. Computer-aided design and manufacturing in craniomaxillofacial surgery: the new state of the art. J Craniofac Surg. 2012 Jan;23(1):288-93. doi: 10.1097/SCS.0b013e318241ba92. PMID 22337427
- [Background] Shiraishi I, Yamagishi M, Hamaoka K, Fukuzawa M, Yagihara T. Simulative operation on congenital heart disease using rubber-like urethane stereolithographic biomodels based on 3D datasets of multislice computed tomography. Eur J Cardiothorac Surg. 2010 Feb;37(2):302-6. doi: 10.1016/j.ejcts.2009.07.046. Epub 2009 Sep 15. PMID 19758813
- [Background] Suarez-Mejias C, Gomez-Ciriza G, Valverde I, Parra Calderon C, Gomez-Cia T. New technologies applied to surgical processes: Virtual Reality and rapid prototyping. Stud Health Technol Inform. 2015;210:669-71. PMID 25991234
- [Background] Valverde I, Gomez G, Gonzalez A, Suarez-Mejias C, Adsuar A, Coserria JF, Uribe S, Gomez-Cia T, Hosseinpour AR. Three-dimensional patient-specific cardiac model for surgical planning in Nikaidoh procedure. Cardiol Young. 2015 Apr;25(4):698-704. doi: 10.1017/S1047951114000742. Epub 2014 May 9. PMID 24809416
- [Background] Valverde I, Gomez G, Coserria JF, Suarez-Mejias C, Uribe S, Sotelo J, Velasco MN, Santos De Soto J, Hosseinpour AR, Gomez-Cia T. 3D printed models for planning endovascular stenting in transverse aortic arch hypoplasia. Catheter Cardiovasc Interv. 2015 May;85(6):1006-12. doi: 10.1002/ccd.25810. Epub 2015 Feb 12. PMID 25557983
- [Background] Valverde I, Gomez-Ciriza G, Hussain T, Suarez-Mejias C, Velasco-Forte MN, Byrne N, Ordonez A, Gonzalez-Calle A, Anderson D, Hazekamp MG, Roest AAW, Rivas-Gonzalez J, Uribe S, El-Rassi I, Simpson J, Miller O, Ruiz E, Zabala I, Mendez A, Manso B, Gallego P, Prada F, Cantinotti M, Ait-Ali L, Merino C, Parry A, Poirier N, Greil G, Razavi R, Gomez-Cia T, Hosseinpour AR. Three-dimensional printed models for surgical planning of complex congenital heart defects: an international multicentre study. Eur J Cardiothorac Surg. 2017 Dec 1;52(6):1139-1148. doi: 10.1093/ejcts/ezx208. PMID 28977423
- [Background] Infante-Cossio P, Prats-Golczer V, Gonzalez-Perez LM, Belmonte-Caro R, Martinez-DE-Fuentes R, Torres-Carranza E, Gacto-Sanchez P, Gomez-Cia T. Treatment of recurrent mandibular ameloblastoma. Exp Ther Med. 2013 Aug;6(2):579-583. doi: 10.3892/etm.2013.1165. Epub 2013 Jun 18. PMID 24137230
- [Background] Hevia V, Ciancio G, Gomez V, Alvarez S, Diez-Nicolas V, Burgos FJ. Surgical technique for the treatment of renal cell carcinoma with inferior vena cava tumor thrombus: tips, tricks and oncological results. Springerplus. 2016 Feb 20;5:132. doi: 10.1186/s40064-016-1825-1. eCollection 2016. PMID 26933631
- [Derived] Rivero Belenchon I, Congregado Ruiz CB, Gomez Ciriza G, Gomez Dos Santos V, Burgos Revilla FJ, Medina Lopez RA. Impact of 3D-Printed Models for Surgical Planning in Renal Cell Carcinoma With Venous Tumor Thrombus: A Randomized Multicenter Clinical Trial. J Urol. 2025 May;213(5):568-580. doi: 10.1097/JU.0000000000004425. Epub 2025 Jan 21. PMID 39836858